CLINICAL TRIAL: NCT07239232
Title: Assessment Of Knee Joint Position Sense And Dynamic Balance IN Female With Primary Dysmenorrhea
Brief Title: "Knee Joint Position Sense and Dynamic Balance in Females With Primary Dysmenorrhea
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Belal Ahmed, Principal Investigator, Cairo University
Other Study IDs: P.T.REC/012/005972
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Primary Dysmenorrhea
Keywords: Knee; Position sense; Balance; Primary Dysmenorrhea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asymptomatic Group: They have no or mild primary dysmenorrhea.
  Interventions: Other: No intervention
- Symptomatic Group: They have moderate and sever primary dysmenorrhea.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of the study is to assess knee joint position sense, pain and dynamic balance in female with primary dysmenorrhea.

DETAILED DESCRIPTION:
Dysmenorrhea is a common condition that typically occurs on its own rather than as a result of pelvic disease. It affects between 50% and 90% of adolescent girls and women of reproductive age and is a major reason for missed days from school or work.

Among the various menstrual disturbances observed, dysmenorrhea was notably prevalent among adolescents and significantly impacted their daily activities. Early diagnosis and awareness of menstrual issues are crucial, as they not only emphasize the need for health education initiatives but also assist in selecting suitable treatments, thereby reducing the adverse effects of these disturbances on adolescents' lives.

However, there is a significant gap in the literature about the effect of Primary dysmenorrhea on knee joint position sense, pain and dynamic balance in young adult female So this study aims to investigate this effect and provide evidence based information in the field of physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* They should be virgin, healthy female students
* They have regular menstruation (3-8 days in duration, with 21-35 days in-between).
* They should have the same activity level mild active female.
* Their ages will range from 18 to 25 years old.
* Their body mass index (BMI) will range from 18 to 24.9 Kg/m2.

Exclusion Criteria:

* History of knee injury, surgery in the knee or spinal vertebrae.
* Females having any vestibular problems, otitis media, labyrinthitis or any inner ear problems that affect balance
* Women with any cognitive deficits
* History of neuromuscular or spinal disease.
* History of pelvic pathology or any gynecological disease.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sixty-two healthy female university students will participate in this study. They will be selected randomly from faculty of physical therapy, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Overall Stability Index (OSI) . Antero-posterior stability index score (APSI) . Medio lateral stability index score (MLSI) . Over all stability index score (OASI) | at first and fourth menstrual days
  The Overall Stability Index (OSI) is the primary measure of dynamic postural control obtained from the balance assessment system. It reflects the standard deviation of the participant's sway from the platform's center across both the medial-lateral and anterior-posterior directions. Higher OSI values indicate greater instability and poorer balance performance. As an integrated measure of sway variability, the OSI is considered the most comprehensive indicator of overall balance ability and is commonly used to evaluate changes in postural control in response to therapeutic interventions.
Medial-Lateral Stability Index (MLSI) | at first and fourth menstrual days
  The Medial-Lateral Stability Index (MLSI) quantifies the degree of side-to-side sway during balance testing. It represents the standard deviation of medial-lateral movement from the platform's center point, providing a directional measure of postural stability. Elevated MLSI scores reflect increased lateral instability, which may be associated with impaired neuromuscular control or deficits in weight-shifting ability. This variable is useful for identifying balance impairments that predominantly affect frontal plane stability.
Anterior-Posterior Stability Index (APSI) | at first and fourth menstrual days
  The Anterior-Posterior Stability Index (APSI) measures front-to-back sway during dynamic balance assessment. Calculated as the standard deviation of anterior-posterior deviations from the center of the platform, the APSI provides insight into sagittal plane stability. Higher APSI values indicate greater instability and reduced capacity to control forward and backward movements. This index is important for evaluating postural control related to gait, stepping, and activities requiring controlled anterior or posterior shifts in the center of gravity.
knee joint position sense | at first and fourth menstrual days
  using active knee position sense test by universal goniometer.

SECONDARY OUTCOMES:
knee joint pain | at first and fourth menstrual days
  It will be assessed using the Visual analog scale (VAS) for all females in both groups. They will score their level of pain from 1-10, with higher scores indicating more severe pain. It is valid and reliable in pain assessment

CONTACTS AND LOCATIONS:
Overall Officials: AFAF M BOTLA, PhD, Study Chair — Assistant Professor, Cairo University; ELHAM s HASSAN, PhD, Study Director — Lecturer, Cairo university
Locations (1):
- Cairo University, Giza, Egypt